CLINICAL TRIAL: NCT03086187
Title: The Effects of a 56day Unilateral Muscular Unloading Intervention With a Novel Device That Allows Normal Ambulation While Reducing Muscle Activation Drastically, on Muscles, Bones and Vessels
Brief Title: The Effects of the Novel Unloading Device "HEPHAISTOS" on Bone, Muscles and Vessels
Acronym: HEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HEP
Record Dates: First submitted 2012-07-31; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Muscle; Atrophy, General
Keywords: weight bearing; muscle unloading; bone loss; arterial adaptation; muscular adaptation
MeSH Terms: conditions — Atrophy; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hephaistos unloading orthosis (Other): Hephaistos unloading orthosis: Calf muscle unloading: The 11 male subjects had to wear a novel orthosis for 8 weeks, which greatly reduces plantarflexor forces during gait.
  Interventions: Device: Hephaistos unloading orthosis

INTERVENTIONS:
Device: Hephaistos unloading orthosis — The Hephaistos unloading orthosis greatly reduces plantarflexor muscle torque and plantarflexor muscle activation during any gait activity.

SUMMARY:
11 healthy men used the HEPHAISTOS unloading orthosis in an ambulatory 8 week intervention study.

It greatly reduces calf muscle forces without reducing ground reaction forces.

DETAILED DESCRIPTION:
The 56day unloading intervention with HEPHAISTOS had the following key objectives:

1. Primary objective: Assessment and evaluation of bone adaptation.
2. Secondary objective: Assessment and evaluation of functional and structural muscular adaptations.
3. Third objective: Assessment and evaluation of functional and structural vascular adaptations.
4. Fourth objective: Assessment and evaluation if the present findings deviate from findings observed in established unloading models.

ELIGIBILITY:
Inclusion Criteria:

* male
* age: 20-45
* BMI: 20-30

Exclusion Criteria:

* smoking
* professional sports men
* diabetes
* rheumatism
* muscle and joint disease
* bone fractures within 12 months prior to the study
* cruciate ligament rupture within 10 years prior to the study
* metal implants
* participation in any other clinical study within 2 months prior to the study haemophilia
* any blood vessel disease
* epilepsy
* claustrophobia
* herniated disk
* cardiac pulse generator
* drug or alcohol abuse
* hyperlipidaemia
* kidney disease
* hyperhomocysteaemia
* hyper/hypouricemia
* hyper/hypocalcaemia
* anaemia
* vitamin d deficit
* chronical back pain
* deficient certificate of good conduct
* achilles tendon injury

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Bone density as measured with pQCT | At baseline and up to 12 months after the immobilization phase
  Change from baseline to 14 days after immobilization phase

SECONDARY OUTCOMES:
Structural and functional parameters of arterial adaptation | At baseline and up to 12 months after the immobilization phase
  Change in intima & media thickness.
Structural and functional parameters of arterial adaptation | At baseline and up to 12 months after the immobilization phase
  Change in arterial diameter
Structural and functional parameters of arterial adaptation | At baseline and up to 12 months after the immobilization phase
  Change in blood flow
Structural and functional parameters of arterial adaptation | At baseline and up to 12 months after the immobilization phase
  Change in flow-mediated dilation

CONTACTS AND LOCATIONS:
Overall Officials: Jörn Rittweger, Prof. Dr., Study Director — German Aerospace Center (DLR)
Locations (1):
- German Aerospace Center, Cologne, North Rine Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Webpage of the German Aerospace Center (DLR) — http://www.dlr.de